CLINICAL TRIAL: NCT07249164
Title: Perioperative Dexmedetomidine and 30-Day Outcomes After Adult Cardiac Surgery: A Real-World Retrospective Cohort Study Using the TriNetX Network
Brief Title: Perioperative Dexmedetomidine and 30-Day Outcomes After Adult Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH114-REC3-181
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Delirium - Postoperative; Cardiac Surgical Procedures; Coronary Artery Bypass Graft (CABG); Valve Surgery; Postoperative Complications
Keywords: Dexmedetomidine; Perioperative Care; Cardiac Surgery; Propensity Score Matching; TriNetX
MeSH Terms: conditions — Emergence Delirium; Postoperative Complications | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perioperative Dexmedetomidine: Adults undergoing first-time CABG or valve surgery with any dexmedetomidine recorded from 24 h before to 48 h after the index surgery on TriNetX; exposure observed in routine care, not assigned by investigators.
  Interventions: Drug: Dexmedetomidine
- No Perioperative Dexmedetomidine: Same surgical cohort with no dexmedetomidine recorded within the -24 to +48 h window; use of dexmedetomidine outside this window allowed; comparison reflects perioperative sedation strategy.
  Interventions: Other: Usual care without perioperative dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Exposure in routine care within -24 to +48 hours of the index cardiac surgery; dose and regimen not protocol-assigned; observational only; exposure captured from medication records and used to define the dexmedetomidine cohort.
  Other Names: Precedex
  Groups: Perioperative Dexmedetomidine
Other: Usual care without perioperative dexmedetomidine — No dexmedetomidine administered within -24 to +48 hours of the index surgery; all other management per routine care; observational comparator; dexmedetomidine use outside this window permitted.
  Groups: No Perioperative Dexmedetomidine

SUMMARY:
This observational study uses de-identified electronic health record data from the TriNetX Global Collaborative Network (2010-01-01 to 2025-07-01) to examine whether perioperative dexmedetomidine (DEX) is associated with 30-day outcomes after adult cardiac surgery. Adults aged 18-100 years undergoing first-time coronary artery bypass grafting or heart valve surgery are included. Exposure is any DEX administration from 24 hours before to 48 hours after the index operation; comparators receive no DEX in this window. The primary outcome is delirium within 30 days. Secondary outcomes are 30-day all-cause mortality, acute kidney injury, pneumonia, sepsis, red blood cell transfusion/major bleeding, myocardial infarction, ischemic stroke/transient ischemic attack, atrial fibrillation, mechanical ventilation >96 hours (days 4-30), and 30-day readmission (days 1-30). No treatments are assigned by investigators and no identifiable information is used. Findings aim to inform perioperative sedation strategies in routine cardiac surgery care.

DETAILED DESCRIPTION:
This is a retrospective cohort study using de-identified data from the TriNetX Global Collaborative Network (2010-01-01 to 2025-07-01). Adults aged 18-100 years undergoing first-time coronary artery bypass grafting or heart valve surgery will be identified. Perioperative exposure is defined as any dexmedetomidine administration from 24 hours before to 48 hours after the index surgery; the comparison cohort consists of patients without dexmedetomidine in this window. Clinical outcomes within 30 days after surgery include delirium as the primary outcome and a range of major postoperative complications and mortality. Propensity scores based on demographics, comorbidities, baseline medications and laboratory tests will be used to match or adjust between exposure groups, with balance assessed using standardized mean differences. Time-to-event analyses will use Cox proportional hazards models and Kaplan-Meier curves, with multiplicity controlled using the Benjamini-Hochberg false discovery rate. All analyses use only de-identified data within the TriNetX platform, with no direct contact with patients or access to identifiers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100 years.
* First-time CABG or heart valve surgery within TriNetX during 2010-01-01 to 2025-07-01.
* ≥90 days pre-operative observable data and a 30-day post-operative window (death ≤30 days counts as complete).
* Index surgery, exposure window (-24 to +48 h), and outcomes identifiable from standardized platform codes/fields.

Exclusion Criteria:

* End-stage renal disease or dialysis within 90 days before index surgery (ICD-10-CM N18.6, Z49, Z99.2).
* Not first-time CABG/valve in the same admission.
* Missing required fields or conflicting records preventing unique case definition.
* Unable to confirm exposure window or outcomes within the platform.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-100 years undergoing first-time CABG or valve surgery in the TriNetX Global Collaborative Network (2010-01-01 to 2025-07-01); de-identified EHR data; exposure defined as perioperative dexmedetomidine -24 to +48 h; comparator without dexmedetomidine in that window.
Sampling Method: Non-Probability Sample
Enrollment: 408153 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Delirium within 30 days | Day 0 through Day 30 after index surgery
  Delirium identified from EHR codes (ICD-10-CM/SNOMED CT). TriNetX "exclude prior to window" enabled; patients with delirium before Day 0 excluded from the risk set. Estimates reported as cumulative incidence and Cox HR with 95% CI.

SECONDARY OUTCOMES:
All-cause mortality within 30 days | Day 0 through Day 30 after index surgery
  Death status from death registry/EHR status flags; exclude-prior-to-window enabled; cumulative incidence and Cox HR.
Acute kidney injury within 30 days | Day 0 through Day 30 after index surgery
  Acute kidney injury by ICD-10-CM/SNOMED CT codes; exclude-prior-to-window; cumulative incidence and Cox HR.
Pneumonia within 30 days | Day 0 through Day 30 after index surgery
  Pneumonia by ICD-10-CM/SNOMED CT; exclude-prior-to-window; cumulative incidence and Cox HR.
Sepsis within 30 days | Day 0 through Day 30 after index surgery
  Sepsis by ICD-10-CM/SNOMED CT; exclude-prior-to-window; cumulative incidence and Cox HR.
Red blood cell transfusion or major haemorrhage within 30 days | Day 0 through Day 30 after index surgery
  Any red blood cell transfusion or major bleeding by CPT/HCPCS and ICD-10-CM/SNOMED CT; exclude-prior-to-window; cumulative incidence and Cox HR.
Myocardial infarction within 30 days | Day 0 through Day 30 after index surgery
  Myocardial infarction by ICD-10-CM/SNOMED CT; exclude-prior-to-window; cumulative incidence and Cox HR.
Ischemic stroke or transient ischemic attack within 30 days | Day 0 through Day 30 after index surgery
  Ischemic stroke/transient ischemic attack by ICD-10-CM/SNOMED CT; exclude-prior-to-window; cumulative incidence and Cox HR.
Atrial fibrillation within 30 days | Day 0 through Day 30 after index surgery
  Atrial fibrillation by ICD-10-CM/SNOMED CT; exclude-prior-to-window; cumulative incidence and Cox HR.
Mechanical ventilation >96 hours | Day 4 through Day 30 after index surgery
  Duration of invasive mechanical ventilation >96 h using ICD-10-PCS/CPT/HCPCS/SNOMED CT; exclude-prior-to-window; cumulative incidence and Cox HR.
30-day readmission | Day 1 through Day 30 after index surgery
  Any all-cause hospital readmission from encounter/admission flags (diagnoses on readmission as coded); exclude-prior-to-window; cumulative incidence and Cox HR.

CONTACTS AND LOCATIONS:
Overall Officials: En-Bo Wu, MD, Principal Investigator — Department of Anesthesiology, China Medical University Hospital, Taichung City, Taiwan
Locations (1):
- China Medical University Hospital, Taichung, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
This retrospective observational study uses de-identified data from the TriNetX Global Collaborative Network. Investigators do not receive identifiable information or re-identification keys. The Data Use Agreement with TriNetX and participating health care organizations prohibits sharing or redistributing line-level individual participant data outside the platform. Only aggregate results and model estimates will be shared (e.g., tables, figures); study documents and analysis code may be provided on reasonable request.

REFERENCES:
- [Background] Caetano da Silva L, Tapioca V, Viana P, Pereira EM, Gibicoski T, Amaral S. Dexmedetomidine for delirium prevention after cardiac surgery: An updated systematic review and meta-analysis with trial sequential analysis. Anaesth Crit Care Pain Med. 2025 Sep;44(5):101578. doi: 10.1016/j.accpm.2025.101578. Epub 2025 Jun 24. PMID 40570954
- [Background] Wang HB, Jia Y, Zhang CB, Zhang L, Li YN, Ding J, Wu X, Zhang Z, Wang JH, Wang Y, Yan FX, Yuan S, Sessler DI. A randomised controlled trial of dexmedetomidine for delirium in adults undergoing heart valve surgery. Anaesthesia. 2023 May;78(5):571-576. doi: 10.1111/anae.15983. Epub 2023 Feb 16. PMID 36794600
- [Background] Poon WH, Ling RR, Yang IX, Luo H, Kofidis T, MacLaren G, Tham C, Teoh KLK, Ramanathan K. Dexmedetomidine for adult cardiac surgery: a systematic review, meta-analysis and trial sequential analysis. Anaesthesia. 2023 Mar;78(3):371-380. doi: 10.1111/anae.15947. Epub 2022 Dec 19. PMID 36535747